CLINICAL TRIAL: NCT02103387
Title: Five Sessions Intervention to Facilitate Adaptation to Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Michael H. Antoni, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20060496; 2R01CA064710 (NIH)
Record Dates: First submitted 2014-03-27; First posted 2014-04-03 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Relaxation Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive Behavioral Training (Experimental): Cognitive Behavioral Training 5 weekly 1.5-hour sessions of group-based cognitive behavioral training
  Interventions: Behavioral: Cognitive Behavioral Training
- Relaxation Training (Experimental): Relaxation Training 5 weekly 1.5-hour sessions of group-based relaxation training
  Interventions: Behavioral: Relaxation Training
- Health Education Control (Active Comparator): Health Education Control 5 weekly 1.5 sessions of group-based health education training
  Interventions: Behavioral: Health Education Control

INTERVENTIONS:
Behavioral: Cognitive Behavioral Training — Cognitive Behavioral Training [CBT] (stress awareness, cognitive restructuring, coping skills training, interpersonal skills training)
  Arms: Cognitive Behavioral Training
Behavioral: Relaxation Training — Relaxation Training [RT] (muscle relaxation, deep breathing, guided imagery, meditation)
  Arms: Relaxation Training
Behavioral: Health Education Control — Health Education control condition (information about breast cancer diagnosis and treatment, side-effect management, recurrence, physical activity and nutrition, and life after breast cancer)
  Arms: Health Education Control

SUMMARY:
To test the effects of 2 different 5-wk stress management interventions (cognitive behavioral training or relaxation training) vs. a time-matched 5-wk health education condition on psychosocial adaptation and physiological adaptation in women being treated for breast cancer. Participants assigned to either of the stress management conditions will show improved psychosocial adaptation and physiological adaptation compared to those assigned to the health education condition.

DETAILED DESCRIPTION:
This is a randomized controlled trial comparing the effects of 5-wk group-based stress management interventions (cognitive behavioral therapy [CBT] or relaxation training [RT]) vs a time-matched 5-wk group-based health education (HE) condition on psychosocial adaptation (negative and positive mood, social disruption) and physiological adaptation (cortisol and immune function) in women with non-metastatic breast cancer who are undergoing primary treatment. Participants are recruited in the weeks after surgery and before the start of adjuvant chemotherapy or radiation, are assessed for baseline psychosocial and physiological adaptation indicators, and are then randomly allocated to either CBT, RT or HE. They are re-assessed for psychosocial and physiological adaptation at 6 and 12 month follow-up. Primary hypothesis is that women assigned to CBT or RT will show greater reductions in negative affect and social disruption, and greater increases in positive affect over time compared to women assigned to HE. Secondary hypothesis is that women assigned to CBT or RT will show greater decreases in cortisol and greater increases in immune functioning over time compared to those assigned to HE.

ELIGIBILITY:
Inclusion Criteria:

* women diagnosed with breast cancer at stage III or below who had recently undergone lumpectomy or mastectomy

Exclusion Criteria:

* prior cancer, prior psychiatric treatment for a serious disorder (e.g., psychosis, suicidality), lack of fluency in English and had begun adjuvant therapy at time of first assessment

Ages: 21 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2007-01-02 (Actual); Primary Completion 2014-02-25 (Actual); Study Completion 2014-02-25 (Actual)

PRIMARY OUTCOMES:
Negative affect as measured by the Affect Balance Scale- Negative Affect subscale | Changes in scores from baseline to 12-month follow-up
  Change from baseline to 12-month follow-up in the Affect Balance Scale- Negative Affect subscale. The Affect Balance Scale includes 40 adjectives assessing negative and positive mood. The Negative Affect subscale (i.e., depression, hostility, guilt, anxiety) will be used. Each emotional state is rated on a Likert Scale (0=never to 5= always) based on the past week and items are averaged, with higher scores indicating more negative affect. Possible scores range from 0-5.
Positive affect as measured by the Affect Balance Scale- Positive Affect subscale | Changes in scores from baseline to 12-month follow-up
  Change from baseline to 12-month follow-up in the Affect Balance Scale- Positive Affect subscale. The Affect Balance Scale includes 40 adjectives assessing negative and positive mood. The Positive Affect subscale (i.e., affection, contentment, vigor, joy) will be used. Each emotional state is rated on a Likert Scale (0=never to 5= always) based on the past week and items are averaged, with higher scores indicating more positive affect. Possible scores range from 0-5.
Social disruption as measure by the Sickness Impact Profile- Social Interaction subscale | Changes in scores from baseline to 12-month follow-up
  Change from baseline to 12-month follow-up in the Sickness Impact Profile- Social Interaction subscale, a 16-item subscale measuring the level of disruption in social activities. Respondents are asked statements regarding social disengagement as they specifically apply to their breast cancer (e.g., "I am doing fewer social activities with groups of people") over the past few weeks, and are asked to respond either No (0) or Yes (1), this applies to me. Scores are summed, with higher scores indicating greater social disruption. Possible scores range from 0-16.

SECONDARY OUTCOMES:
Physiological Adaptation | 12 month follow-up
  Change from baseline to 12 month follow-up in physiological adaptation (decreased serum cortisol, and increased Th1 cytokine production and lower Th2 cytokine production following anti-CD3 stimulation of peripheral blood mononuclear cells (PBMCs)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Antoni, Ph.D., Principal Investigator — University of Miami
Locations (1):
- Department of Psychology, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ream M, Saez-Clarke E, Taub C, Diaz A, Frasca D, Blomberg BB, Antoni MH. Brief Post-Surgical Stress Management Reduces Pro-Inflammatory Cytokines in Overweight and Obese Breast Cancer Patients Undergoing Primary Treatment. Front Biosci (Landmark Ed). 2022 May 7;27(5):148. doi: 10.31083/j.fbl2705148. PMID 35638415
- [Derived] Diaz A, Taub CJ, Lippman ME, Antoni MH, Blomberg BB. Effects of brief stress management interventions on distress and leukocyte nuclear factor kappa B expression during primary treatment for breast cancer: A randomized trial. Psychoneuroendocrinology. 2021 Apr;126:105163. doi: 10.1016/j.psyneuen.2021.105163. Epub 2021 Feb 4. PMID 33611132